CLINICAL TRIAL: NCT05533606
Title: Analysis of Risk Factors of Beta-Lactam Drugs Related Acute Kidney Injury in Hospitalized Patients and Developments of Machine Learning Model
Brief Title: Risk Factors and Machine Learning Model for Beta-Lactam Drugs Related Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: LCYY-LX-20220103
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury; Beta-Lactam Antibiotic Toxicity (Diagnosis)
Keywords: Beta-Lactam drugs; Acute kidney injury; Pharmacoepidemiology; Miss diagnosis; Risk factors; Logic regression
MeSH Terms: conditions — Acute Kidney Injury; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group
  Interventions: Drug: Beta-Lactam Drugs
- Non-AKI Group
  Interventions: Drug: Beta-Lactam Drugs

INTERVENTIONS:
Drug: Beta-Lactam Drugs — During hospitalization，patients used Beta-Lactam drugs.

SUMMARY:
Acute kidney injury (AKI), also known as acute kidney failure (ARF), is a common and complex kidney disease in clinic and an important factor related to poor prognosis of patients in clinic. In the present study, a single-center retrospective study was conducted in our center. The clinical data of hospitalized patients received β-Lactam drugs from January 2018 to December 2020 was retrospectively analyzed. The multiple logistic regression analysis suggested that complicated with hypertension, anemia, pneumonia, shock, sepsis, heart failure, combined use of proton pump inhibitors (PPI), angiotensin-converting enzyme inhibitor (ACEI), angiotensin Ⅱ receptor antagonist (ARB) were independent risk factors for AKI related to β-Lactam drugs. In clinical practice, patients with acute kidney injury risk factors should be closely monitored for changes in their blood creatinine and urine output to avoid acute kidney injury. For patients who have suffered from acute kidney injury, the cause should be removed in time and corresponding symptomatic treatment should be given.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients who used β-lactam drugs during hospitalization
* Hospital stay ≥ 48h
* Age ≥18 years
* There are two or more blood creatinine tests during hospitalization

Exclusion Criteria:

* Hospital stay < 48h
* Age <18 years
* Glomerular filtration rate (GFR)< 30ml/min/1.73m2 within 48 hours after admission
* AKI was diagnosed on admission
* Less than two Scr test results during hospitalization
* The Scr values were always lower than 40 μmol/L during hospitalization
* Cases with incomplete medical history information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were included if received treatment with β-lactam drugs and discharged from the hospital between January 1, 2018 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of acute kidney injury in hospitalized patients treated with β-lactam drugs | Through study completion，up to half a year.
  To analyze the incidence of acute kidney injury in hospitalized patients after using β-lactam drugs and to build a prediction model.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li，MD, Jinan, Shandong, China